CLINICAL TRIAL: NCT03360708
Title: Pilot Clinical Trial of Allogeneic Tumor Lysate-Pulsed Autologous Dendritic Cell Vaccination in Recurrent Glioblastoma
Brief Title: Vaccine Therapy in Treating Patients With Recurrent Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1772; NCI-2017-02159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1772 (Other: Mayo Clinic)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Giant Cell Glioblastoma; Recurrent Glioblastoma; Recurrent Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on days 1, 3, and 5 of courses 2 and 3, and on day 1 of subsequent courses. Treatment with malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine repeats every 21 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Malignant Glioma Tumor Lysate-Pulsed Autologous Dendritic Cell Vaccine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Malignant Glioma Tumor Lysate-Pulsed Autologous Dendritic Cell Vaccine — Given ID

SUMMARY:
This pilot early phase I trial studies the side effects of vaccine therapy in treating patients with glioblastoma that has come back. Vaccines made from a person's white blood cells mixed with tumor proteins from another person's glioblastoma tumors may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy may work better in treating patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine (autologous dendritic cell [DC] / allogeneic glioblastoma multiforme [GBM] culture lysate vaccination) in glioblastoma patients at first or second recurrence.

SECONDARY OBJECTIVES:

I. To document survival and progression-free survival in glioblastoma patients at first or second recurrence receiving autologous DC / allogeneic GBM culture lysate vaccination and compared to historical data.

TERTIARY OBJECTIVES:

I. Determine the ability of autologous DC / GBM culture lysate vaccination to generate multiple tumor-associated antigen (TAA)-specific immune responses in GBM patients at first or second recurrence.

II. Assess the relationship between ability tumor induced TAA-specific immune responses and evidence of immunosuppression (peripheral blood immunophenotyping by flow cytometry) following autologous DC / allogeneic GBM culture lysate vaccination in GBM patients at first or second recurrence.

III. Assess the relationship between efficacy endpoints (survival, progression-free survival, tumor response) and tumor-associated antigen immune response following autologous DC / allogeneic GBM culture lysate vaccination

IV. Assess the relationship between efficacy endpoints (survival, progression-free survival, tumor response) and evidence of immunosuppression at baseline and over time with autologous DC / allogeneic GBM culture lysate vaccination.

OUTLINE:

Patients receive malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine intradermally (ID) on days 1, 3, and 5 of courses 2 and 3, and on day 1 of subsequent courses. Treatment with malignant glioma tumor lysate-pulsed autologous dendritic cell vaccine repeats every 21 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* First or second recurrence of previously histologically confirmed glioblastoma (grade 4 astrocytoma)

  * NOTE: gliosarcomas and other grade 4 astrocytoma variants (e.g., giant cell) may be included, primitive neuroectodermal tumor (PNET) variants are excluded; grade 4 oligodendrogliomas or oligoastrocytomas are specifically excluded
* Prior craniotomy and gross total or sub-total resection of tumor at this recurrence NOTE: biopsy of this recurrence alone without attempt at resection does not meet this inclusion criteria (i.e. craniotomy and resection is still required).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/uL
* Monocytes >= 300/uL
* Platelets (PLT) >= 100,000/uL
* Hemoglobin (HgB) >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN
* Creatinine =< 1.5 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Ability to understand and willingness to sign written informed consent
* Willing to return to Mayo Clinic in Rochester, Minnesota for follow-up
* Willing to provide tissue and blood samples for mandatory correlative research purposes
* Fixed or decreasing dose of corticosteroids (or no corticosteroids) >= 7 days prior to registration

Exclusion Criteria:

* Prior treatment

  * Current or prior treatment for this cancer with immunotherapy and/or any other investigational agents
  * Surgery =< 2 weeks prior to registration
  * Radiotherapy =< 12 weeks prior to registration
  * Treatment with bevacizumab or any cytotoxic chemotherapy =< 8 weeks prior to registration
* Any of the following

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV), human T-cell lymphotropic virus (HTLV), hepatitis B (HepB), or hepatitis C (HepC) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of other malignancy other than glioma

  * EXCEPTIONS: non-melanotic skin cancer, carcinoma-in-situ of the cervix, or systemic cancer that has been in documented remission for > 10 years
  * NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 180 days (6 months), or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Active infection =< 5 days prior to registration or fever >/= 38 degrees Celsius (C) within 5 days prior to registration
* History of tuberculosis or positive purified protein derivative (PPD) test
* Inability or unwillingness to have magnetic resonance imaging (MRI) scans performed (e.g. cardiac pacemaker-dependent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11-27 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Incidence of significant toxicity, defined as a dose limiting toxicity (DLT) that is possibly, probably, or definitely related to treatment as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 5 years
  Incidence of significant toxicity will be estimated by the number of patients with significant toxicity divided by the total number of evaluable patients.

SECONDARY OUTCOMES:
Clinical benefit rate | Up to 5 years
  The clinical benefit rate will be estimated by the number of patients with an overall survival for at least 6 months after enrollment or an objective status of CR or PR at any time divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true clinical benefit rate will be calculated.
Duration of response | Date at which the patient?s objective status is first noted to be either a CR or PR to the earliest date progression is documented, assessed up to 5 years
  Duration of response will be summarized descriptively.
Feasibility | Up to 5 years
  The feasibility of the regimen will be estimated by the number of patients who received at least one dose of dendritic cell (DC) injection divided by the total number of patients who received leukapheresis in that arm.
Overall response rate | Up to 5 years
  The overall response rate will be estimated by the number of patients with an objective status of complete response (CR) or partial response (PR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Overall survival | Time from study registration to progression and death due to any cause, assessed up to 5 years
Progression-free survival | Time from study registration to progression and death due to any cause, assessed up to 5 years
Time to response | Date of initiation of vaccination treatment to the date at which the patient?s objective status is first noted to be either a CR or PR, assessed up to 5 years
  Time to response will be summarized descriptively.

OTHER OUTCOMES:
Change in immunologic correlates | Baseline up to 5 years
  Change in immunologic correlates before and after vaccination treatment will be evaluated and summarized both quantitatively and graphically. Will use Spearman rank correlation coefficient to assess the correlations between baseline levels as well as between changes before and after treatment in these immunologic markers. In addition, these immunologic markers will be correlated with cancer and treatment-related outcomes (e.g. response, toxicities). Relationships will also be explored graphically using scatter plots.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Parney, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States